CLINICAL TRIAL: NCT00438139
Title: Phase 1, Pilot Study to Examine the Cardiovascular Effects of Smoked Marijuana, Interactions With Oral Dronabinol, and Effects of Dronabinol on Withdrawal in Marijuana Dependent Volunteers
Brief Title: Ph1 Marinol Interaction Study - Part 1 - 1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Liza Gorgon, NIDA
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-CPU-0011-1
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2007-02

CONDITIONS: Marijuana Dependence
Keywords: marijuana dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

INTERVENTIONS:
Drug: Dronabinol

SUMMARY:
The purpose of this study is to examine the effects of oral dronabinol tetrahydrocannabinol (THC) on withdrawal symptoms in marijuana dependent volunteers, and evaluate the safety, pharmacokinetics (PK), and cardiovascular effects of the combination of oral dronabinol and smoked marijuana to determine if there are potential significant interactions before conducting outpatient studies.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 to 45 years of age
* Must be in good general health
* Must meet DSM-IV criteria for marijuana dependence and are non- treatment seekers at the time of study
* Must be able to provide written informed consent
* Must be able to provide 1 marijuana positive urine specimen (> 50 ng/mL) within the 28-day screening period
* If female and of child bearing potential, must agree to use birth control.

Exclusion

Criteria:

* Please contact site for more information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6
Dates: Start 2007-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular responses

CONTACTS AND LOCATIONS:
Overall Officials: Louis Cantilena, M.D., Principal Investigator — Uniformed Services University of Health Science
Locations (1):
- Uniformed Services University of Health Science, Bethesda, Maryland, United States